CLINICAL TRIAL: NCT04988802
Title: The Effect of Dietary Supplements for Pregnant Women on Levothyroxine Absorption
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Dubrava (Other)
Responsible Party: Principal Investigator, Tomo Lucijanic, Principal Investigator, University Hospital Dubrava
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: ZG2712TL
Record Dates: First submitted 2021-07-25; First posted 2021-08-04 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Hypothyroidism Primary
Keywords: nutritional supplements; levothyroxine; pregnancy; safety
MeSH Terms: conditions — Hypothyroidism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients taking food supplement with levothyroxine (Active Comparator): Patients will start taking food supplement with levothyroxine in the evening, and the other tablet of the food supplement in the evening for 8 weeks.
  Interventions: Dietary Supplement: Prenatal Nutrients Solgar
- Patients taking placebo with levothyroxine (Placebo Comparator): Patients will start taking placebo with levothyroxine in the evening, and the other tablet of the placebo in the evening for 8 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Prenatal Nutrients Solgar — Patients will take dietary supplement Prenatal Nutrients from Solgar
  Arms: Patients taking food supplement with levothyroxine
Other: Placebo — Placebo capsules based on starch.
  Arms: Patients taking placebo with levothyroxine

SUMMARY:
Hypothyroidism is a common disease that is successfully treated with the replacement of thyroid hormones in the form of levothyroxine. Levothyroxine is drug used in the first line of substitution therapy because it appropriately mimics physiological secretion of thyroxine (T4) and its peripheral conversion to triiodothyronine (T3). However, due to its narrow therapeutic index, and because it is administered at very low doses (micrograms - μg), it is particularly sensitive to the absorption phase interactions, which are due to its narrow therapeutic index, mainly clinically significant. In pregnancy, one of the goals is to maintain the values of thyroid stimulating hormone (TSH) in the lower part of the reference interval (below 2,5 milli-International units - mIU/L) for a proper child development. Also, due to increased nutritional needs during pregnancy, nutritional supplements are commonly used by pregnant women on their own initiative, but also often recommended by healthcare personnel. Reviewing the literature, we did not find high quality evidence to suggest the existence or to refute the interaction between dietary supplements for pregnant women and the absorption of levothyroxine. The aim of this study is to investigate this potential interaction between dietary supplements used in pregnancy and levothyroxine absorption in order to test the safety of the use of these preparations in pregnant women who are on replacement therapy with levothyroxine.

DETAILED DESCRIPTION:
Hypothyroidism is a common disease that is successfully treated with the replacement of thyroid hormones in the form of levothyroxine. Levothyroxine is drug used in the first line of substitution therapy because it appropriately mimics physiological secretion of thyroxine (T4) and its peripheral conversion to triiodothyronine (T3). However, due to its narrow therapeutic index, and because it is administered at very low doses (μg), it is particularly sensitive to the absorption phase interactions, which are due to its narrow therapeutic index, mainly clinically significant. In pregnancy, one of the goals is to maintain the values of thyroid stimulating hormone (TSH) in the lower part of the reference interval (below 2,5 mIU/L) for a proper child development. Also, due to increased nutritional needs during pregnancy, nutritional supplements are commonly used by pregnant women on their own initiative, but also often recommended by healthcare personnel. Reviewing the literature, we did not find high quality evidence to suggest the existence or to refute the interaction between dietary supplements for pregnant women and the absorption of levothyroxine. The aim of this study is to investigate this potential interaction between dietary supplements used in pregnancy and levothyroxine absorption in order to test the safety of the use of these preparations in pregnant women who are on replacement therapy with levothyroxine.

Primary goal is to asses if taking of the food supplement for pregnant women with levothyroxine diminishes the absorption of levothyroxine, which is measured through values of TSH, FT4 and FT3.

Secondary and other objectives are to determine whether the use of dietary supplements intended for pregnant women, due to its mineral-vitamin composition, can affect body weight, waist circumference and lipogram values of patients diagnosed with primary hypothyroidism.

This is a prospective randomized double-blind placebo-controlled clinical trial.

The study would include subjects diagnosed with primary hypothyroidism over the age of 18 and on stable LT4 therapy for at least 6 months. Although the study is intended to examine dietary supplements for pregnant women, the said population will be excluded from the study for safety reasons. Given that the mechanism of the vast majority of LT4 interactions is based on the adsorption of levothyroxine on the interfering substance, we believe that potential differences in LT4 absorption between pregnant women and the study population should not affect the clinical interpretation of the results of this study.

Also, patients with thyroid cancer as well as patients at high cardiovascular risk will be excluded from the study. Patients with proven lactose intolerance will also not participate in this study. Patients with proven celiac disease and Giardia Lamblia infection will be excluded from the study. Also, patients diagnosed with atrophic gastritis or H. pylori infection will be excluded from the study. Although the evidence for the effect of bariatric surgery on LT4 absorption is not entirely clear, this group will not be included in the study due to the potential hazard of the effect of said surgery on absorption.

According to the calculated required sample size, for 90% strength of the study, it will be necessary to include at least 37 patients to determine clinically significant interference of these preparations with LT4 absorption. Analysis of the required sample size is shown later.

Upon entering the study, patients would undergo a medical examination to examine satisfactory inclusive and exclusion criteria for the study, blood sampling for TSH, FT3, FT4, total and ionized calcium, iron, UIBC, TIBC, ferritin, folic acid, vitamin B12, KKS , total cholesterol, HDL, LDL, triglycerides, as well as by measuring anthropometric variables such as body height, body weight, and waist circumference. Waist circumference will be measured according to WHO recommendation at a point located between the lower edge of the lowest palpable rib and the lateral ridge (iliac crest) using a non-extensible measuring tape at the end of normal exhalation in two consecutive measurements. Upon inclusion, subjects will be informed of the study, including that changes in TSH, FT3, and FT4 levels are possible and that they report to the study leader if they experience any disturbances. The study will also be discontinued, subject blindness, and therapy corrected if TSH is greater than or equal to 10mIU / L.

After inclusion, patients will be randomized into two groups in a 1: 1 ratio - one group will take the selected dietary supplement for pregnant women for 8 weeks at the same time as LT4 which will be taken according to the method recommended in the Summary of Product Characteristics-SmPC (half an hour before breakfast with a glass of water), while the second tablet of the preparation intended for pregnant women will be taken in the evening - 12 hours after the morning dose (29). The second group of subjects will take a placebo tablet whose composition will be based on starch. The selected dietary supplement for pregnant women is Prenatal nutrients from Solgar. The preparation was selected from several other preparations based on the widespread use in the pregnant population of our region and beyond.

Randomization as well as the procedure in which the study will be blinded for the involved doctors, but also patients, will be performed in a pharmacy under the supervision of a pharmacist.

It is important to emphasize that when entering the study, patients will be informed about the influence of certain foods (dietary fiber, soy, coffee, grapefruit, vitamin C) on the absorption of LT4 (28). Because these interactions can be avoided by separating the intake of these foods and LT4, patients will be informed by the physician who included them in the study upon entering the study. They will also complete a questionnaire during study entry as well as during follow-up examinations to check their eating habits related to foods that may have an impact on LT4 absorption.

After 8 weeks, a control examination will be performed, during which a blood sample will be taken to determine thyroid hormones and other findings, as well as when included in the study, the aforementioned anthropometric variables will be checked and the doctor will perform examinations to evaluate patient safety. Subsequently, patients who were randomized to the group taking LT4 with dietary supplementation will continue to take LT4 along with placebo, while patients who took LT4 with placebo will continue to take LT4 along with dietary supplement intended for pregnant women. At the end of the second part of the study, a blood sample will be taken again, the examined anthropometric variables will be checked, and the patient will leave the study and continue to take LT4 according to the usual way of taking it.

The study used a period of 8 weeks for each intake regimen as it is a time period that has been proven in several studies to be sufficient to determine changes in LT4 absorption at TSH values (10,11).

Lipidogram values will be measured due to literature data suggesting a beneficial effect of biotin on lipid values, and in the test preparation biotin is present in a dose higher than the recommended daily dose (30, 31, 32, 33).

Upon entering the study, patients will fill out an informed consent in which they will be explained the purpose, procedures and duration of the study. At the time of enrollment in the study and at the end of each observed period of 8 weeks, patients would have a blood sample taken to examine the required parameters.

FT4 and fT3 concentrations will be measured by radioimmunochemical methods, TSH values by immunochemical methods, while anthropometric measurements of body height and weight and waist circumference will be made using calibrated measuring instruments. Determining the values of the required laboratory parameters as well as taking samples will be done according to the standard protocols of the Clinical Institute for Laboratory Diagnostics at the Clinical Hospital Dubrava.

A randomization scheme will be generated at http://www.randomization.com. Patients will be randomized to a dietary supplement intended for pregnant women or placebo, and after 8 weeks of the study will cross-replace the active preparation with placebo and vice versa.

The required number of 37 subjects was obtained using a t-test for paired samples (MedCalc ver. 18.11.6), error type 1 of 0.05, error type 2 of 0.1 (90% strength), standard deviation of differences of 1, 81 and a clinically significant difference in TSH between the two groups of 1.0 mIU / L (11,12). A similar number of subjects were included in earlier studies by other authors that showed the influence of certain substances in the diet on LT4 absorption (13-16, 18).

The normality of the distribution of numerical variables will be tested by the Shapiro-Wilk test. Normally distributed numerical variables will be presented as the arithmetic mean ± standard deviation, and a t-test for paired samples will be used to compare them between the active preparation and the placebo. Non-normally distributed numerical variables will be presented as median and interquartile range, and the Wilcoxon pairwise test will be used to compare them between the active preparation and the placebo. The category variables will be presented as a ratio and a percentage and will be compared between the active preparation and the placebo by the McNemar test. The t-test or Mann Whitney U test for numerical variables, depending on the normality of their distribution, and the χ2 test or Fisher's test for categorical variables will be used to compare patient characteristics at the beginning of the study and parameters of interest at individual time points during the study. P values <0.05 will be considered statistically significant. The MedCalc statistical program (MedCalc Statistical Software version 18.11.6 or later; MedCalc Software bvba, Ostend, Belgium) / licensed to Marko Lucijanić will be used for all analyzes.

ELIGIBILITY:
Inclusion Criteria:

* female patients older than 18 on stable levothyroxine therapy for at least 6 months

Exclusion Criteria:

* Pregnancy
* thyroid carcinoma
* high cardiovascular risk
* coeliac disease
* Giardia Lamblia infection
* atrophic gastritis
* Helicobacter pylori infection
* previous bariatric surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2021-10-20 (Estimated); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in thyrothropin | 8 weeks
  Change in thyrothropin larger than 1mIU/L

CONTACTS AND LOCATIONS:
Locations (1):
- Dubrava University Hospital, Zagreb, City of Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers.

REFERENCES:
- [Background] Fish LH, Schwartz HL, Cavanaugh J, Steffes MW, Bantle JP, Oppenheimer JH. Replacement dose, metabolism, and bioavailability of levothyroxine in the treatment of hypothyroidism. Role of triiodothyronine in pituitary feedback in humans. N Engl J Med. 1987 Mar 26;316(13):764-70. doi: 10.1056/NEJM198703263161302. PMID 3821822
- [Background] Mandel SJ, Brent GA, Larsen PR. Levothyroxine therapy in patients with thyroid disease. Ann Intern Med. 1993 Sep 15;119(6):492-502. doi: 10.7326/0003-4819-119-6-199309150-00009. PMID 8357116
- [Background] Toft AD. Thyroxine therapy. N Engl J Med. 1994 Jul 21;331(3):174-80. doi: 10.1056/NEJM199407213310307. PMID 8008032
- [Background] Wiersinga WM. Thyroid hormone replacement therapy. Horm Res. 2001;56 Suppl 1:74-81. doi: 10.1159/000048140. PMID 11786691
- [Background] Kabadi UM, Jackson T. Serum thyrotropin in primary hypothyroidism. A possible predictor of optimal daily levothyroxine dose in primary hypothyroidism. Arch Intern Med. 1995 May 22;155(10):1046-8. PMID 7748047
- [Background] Helfand M, Crapo LM. Monitoring therapy in patients taking levothyroxine. Ann Intern Med. 1990 Sep 15;113(6):450-4. doi: 10.7326/0003-4819-113-6-450. PMID 2143640
- [Background] Vrhovac i sur. Interna medicina. 3. izdanje. Medicinska biblioteka; 2003. str.1242-1244.